CLINICAL TRIAL: NCT06191653
Title: The Efficacy of a Mindful Self-compassion Based Program With Caregivers of Young Offenders Placed at the Portuguese Juvenile Justice Facilities
Brief Title: Mindfulness and Self-Compassion With Caregivers Working With Delinquent Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Marlene Cristina Mourato Paulo, Principal Investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.06452.BD
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Caregivers of Delinquent Youth
Keywords: Caregivers; Clinical Trial; Delinquent youth; Mindful Self-Compassion
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This project will use a longitudinal design. Caregivers recruited from 4 (out of 6) YDC, selected based the number of available caregivers, were allocated to two conditions: 2 to the treatment group and the other 2 to the wait-list control group. The criteria of this allocation was the number of caregivers available in each institution: the treatment group was composed of the two YDC with the larger number of caregivers in order to increase the chance of having a greater number of participants and dealing with natural dropout levels. A sample of youth was all recruited in all 4 YDC to assess the indirect impact of the intervention program. This trial included a Treatment group (N=34), a Waiting list Control group (N=36), and a sample of youth (45 recruited from the Treatment YDC and 31 recruited from the Control YDC).
Who Masked: Outcomes Assessor
Masking Description: This project will use a longitudinal design. Caregivers recruited from 4 (out of 6) YDC, selected based the number of available caregivers, will be allocated to two conditions: 2 to the treatment group and the other 2 to the wait-list control group. The criteria of this allocation is the number of caregivers available in each institution: the treatment group will be composed of the two YDC with the larger number of caregivers in order to increase the chance of having a greater number of participants and dealing with natural dropout levels. A sample of youth will be recruited in all 4 YDC to assess the indirect impact of the intervention program. This trial will include a Treatment group (N=25), a Waiting list Control group (N=25), and a sample of youth (20 recruited from the Treatment YDC and 20 recruited from the Control YDC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): The adapted form of the MSC, composed for 12 sessions, will be delivered on a weekly basis in group. This intervention program intends to cultivate a compassionate-self as well as increase the awareness of personal patterns of functioning and learning to respond to them in a kind, courageous, and fierce way. All the sessions will be delivered in a space on each YDC.
  Interventions: Behavioral: Mindfulness and Self-Compassion for Caregivers working in Youth Detention Centres
- Control Group (No Intervention): This group, wich will be a waiting list control goup, will not receive any mind training or group intervention during the study. Participants of this group will be assessed at 4 different time points (pre- and post-treatment and at a 3- and 6-month follow-up). After all assessment moments are completed, the intervention program will be delivered with the caregivers of this group. These caregivers will receive the intervention after the end of all assessment moments and at a time to be agreed with the Portuguese Juvenile Ministry of Justice. Adolescents cared both by wokers in the TG and CG will not receive any intervention during the study.

INTERVENTIONS:
Behavioral: Mindfulness and Self-Compassion for Caregivers working in Youth Detention Centres — The adapted form of the MSC is a 12-session structured program, delivered on a weekly basis in group. It intends to cultivate a compassionate-self as well as increase the awareness of personal patterns of functioning and learning to respond to them in a kind and courageous way. Each session lasts about 2 hours. Each session has the following structure: Grounding exercise; sharing individual insights about the weekly practice; Reviewing the previous session and link for the session theme; coffee break; soft landing exercise; Formal/Informal practice(s); Session summary and challenges to be applied during the week; Session evaluation and take-off. Each participant receives a manual with the contents shared in each session as well as some space for individual reflections. On the day after each session, a summary email is sent to the participants, resuming the contents and with records of the (in)formal practices delivered. All the sessions will be delivered in a space on each YDC.
  Arms: Treatment group

SUMMARY:
The work carried out in Youth Detention Centers (YDC) represents a set of challenges for caregivers, who are in the frontline of juvenile delinquency. These professionals have daily to cope daily with work and relational challenges, while experiencing high levels of stress and physical and emotional fatigue. As such, taking care of the well-being of these professionals is of paramount importance, moreso as they are fundamental in the rehabilitation of young offenders. Still, the usual training/interventions offered to these professionals does not consider/fit to their psychological, emotional, or psychical difficulties. Recent studies have explored the impact of contextual cognitive-behavioral interventions with caregivers (e.g., parents of individuals with developmental disabilities, nurses, healthcare providers), namely those based on Mindfulness and Self-Compassion. The Mindfulness Self-Compassion Program (MSC) has been found to be effective in reducing caregivers' overwhelmed feelings about their own suffering and/or the suffering of others.

This clinical trial intends to explore the adequacy of the adapted form of MSC (12 group sessions) to caregivers working in YDC, and to establish its effectiveness. Two main studies will be carried out: 1) a parallel non-randomized clinical trial, in which the effectiveness of the program will be explored, as well as the mechanisms of change of the participants' responsiveness to the intervention; and 2) individual interviews to assess qualitatively the participants' perception about the usefulness and impact of the intervention (concerning their relationship with youth and with work colleagues, their relationship with themselves and the general climate of the YDC). A sample of youth placed in each selected YDC will be recruited and will be assessed through self-report questionnaires at the same moments as caregivers samples. It is hypothesized that the adapted form of MSC will produce significant improvements in outcome measures when comparing caregivers who receive the intervention program with those in the control group. Specifically, it is expected an improvement in caregivers' positive feelings and well-being, in their sensitivity and compassion towards others' suffering, as well as a decrease on some indicators of stress and suffering. Consequently, it is also expected that youth in YDC perceive more warmth and safeness experiences with caregivers and report increases in their interpersonal functioning.

DETAILED DESCRIPTION:
Youth delinquency is a relevant social problem and there is growing interest in improving intervention with young offenders. Interventions developed at the Youth Detention Centers (YDC) involve several human resources, who daily supervise the youth routines, care for them, and model their behaviors. The challenges and difficulties of working with people with delinquent behavior have been explored in different groups of caregivers, but little studied in caregivers of young offenders. Such difficulties are identified as risk factors for the development of physical and psychological symptoms in caregivers, and seem to be related to personal issues (e.g., gender, age, education level, personal beliefs, work-related motivations and levels of perceived social support), but also with issues inherent to the work context, characterized as challenging, demanding and of great responsibility (e.g., the ambiguity of professional role, time spent in a corrective context, supervision, and support from hierarchical superiors, job satisfaction, and commitment. Some authors argue that the constraints placed on caregivers significantly predict high levels of stress and compassion fatigue/burnout manifested by symptoms of depression, anxiety, and physical/psychological exhaustion, with a negative impact on levels of compassion for others, on the performance of professional duties and on the satisfaction of those who are cared for. As a result of these difficulties, self-care practices have been recommended in order to prevent and/or relieve these symptoms in caregivers. Still, also in Portugal, tutelary/educative interventions are predominant, with efforts being focused on the psychological rehabilitation of delinquent youth and disregarding those responsible for that rehabilitation.

Recent research has evaluated the impact of contextual cognitive-behavioral interventions with groups of caregivers. Interventions based on Mindfulness, which aims to promote non-reactive awareness of thoughts, emotions, and bodily sensations, and those that promote Self-compassion have stood out for their effectiveness. In particular, the Mindful Self-Compassion Program (MSC) encompasses the two previously described components and, despite being less studied than approaches based solely on Mindfulness, has gathered effectiveness evidence with various groups of caregivers (e.g., nurses, healthcare providers) and on skills considered essential for caregivers to respond to the needs of those they care (e.g., reduction of physical/psychological problems; increases quality/satisfaction with life and levels of empathy and compassion towards others. Recent research has shown that the MSC seems to be effective in reducing the caregiver's feeling of burden with their own suffering and/or with the suffering of others.

Despite the importance of establishing positive and safe relationships between young offenders and their caregivers, studies carried out with caregivers are scarce and focus mainly on assessing their needs and/or difficulties, not aiming to intervene on them. Interventions offered to these caregivers aim to train them to deal with youth behavioral problems, to improve their knowledge on delinquent developmental trajectories, or to improve the physical/relational settings of caregiving contexts.

This work aims to fulfill this gap, by studying the effectiveness of an adapted form of MSC in promoting self-care and satisfaction with life and work, which are considered essential for effective care provision, in caregivers of young people in Portuguese YDC. This clinical trial is a parallel non-randomized controlled trial, designed according to the CONSORT guidelines, and carried out in 4 (out of 6) YDC. It aimed to test the efficacy of an adapted form of the MSC applied to caregivers working on YDC. It is expected that the application of the adapted form of MSC to the YDC caregivers will contribute to an increase in caregivers' physical, emotional, and psychological well-being and job satisfaction. In addition, it is also expected that the improvements mentioned above have a positive impact on the quality of the provided care and the interpersonal functioning of delinquent youth.

All procedures involved in this project (described elsewhere in this form) were carried out according to the ethical principles of the Declaration of Helsinki and the applicable national laws and regulations. Moreover, all procedures were approved by the Ethics Committee of the Faculty of Psychology and Educational Sciences, University of Coimbra as well as by the Portuguese Juvenile Ministry of Justice.

Informed consent will be required for all potential participants prior to any data collection. Caregivers will give informed consent. Adolescents aged between 14 and 16 years old (YO), will give informed assent, while those older than 16 YO will give written informed consent. A written informed consent will be gathered from guardians/legal representatives of all adolescent participants under 18 YO. All participants (i.e., caregivers and adolescents, as well as their parents/legal guardians) will be informed that their participation is voluntary and that they could decline to participate at any time during the project without any negative consequence. Moreover, participants will be informed that the confidentiality of responses would be assured at all moments. The anonymity of all participants' responses is guaranteed, with the use of respondent-specific codes, which will be also used to link the data from one time point to the other.

From the 6 Portuguese YDC, 4 will be selected considering the number of caregivers. YDC with the highest number of staff will be selected for participation. Two YDC will be allocated to the Treatment Group (TG) and the other two to the Control Group (CG); one treatment and one control group will be considered during the year of execution of this research, and the other treatment and control groups will be sequentially considered in the following year after all procedures with the first groups were concluded.

Caregivers in the TG will attend the adapted form of MSC for about 12 weeks. The intervention consists of 12 two-hour weekly group sessions (including a 10-minute coffee break), delivered in each YDC to a group of 4 to 8 participants. The hours spent participating in the project (24 hours) will be given as time off. Caregivers in the CG, which functions as a waiting list control group, did not receive any intervention during the study. It is intended that those caregivers receive the intervention after the end of all assessment moments and at a time to be agreed with the Portuguese Juvenile Ministry of Justice. Adolescents cared both by workers in the TG and CG will not receive any intervention during the study. Treatment integrity will be ensured through: a) specific treatment manuals; b) direct training of the therapist and c) supervision by a senior therapist, with advanced training on the MSC program.

Caregivers of both groups will fill out the assessment protocol individually during working hours in each YDC and the adolescents of both groups will complete the self-report questionnaires, individually, in the presence of the researcher responsible for the project. All participants (caregivers and adolescents) will be assessed through self-report measures 4 times across 12 months. Specifically, participants will be assessed before the first session of the program (baseline - time 1), right after its terminus (i.e., post-treatment assessment - time 2), and 3 and 6 months after intervention terminus (follow-up 1 and 2 - time 3 and time 4). Participants in the control group (both youth and caregivers) will be assessed using the same self-report instruments and with the same time intervals as those in the intervention group. Quantitative analyses will be carried out according to the principle of Intention-to-treat analysis (including all participants regardless of whether or not they participated in all sessions). Analyses will also be carried out only with participants who completed the protocol (Peer-protocol analysis). Treatment effects and covariate effects will be analysed with mixed MANOVAs. Change mechanism studies will be analysed with two-wave latent growth curve models.

On 3 and 6-months follow-up assessments, in addition to the assessment protocol, caregivers of the TG will also be qualitatively evaluated, through individual interviews. The participants will be asked about their perception of the impact of participating in the MSC program on their relationships at the YDC (namely with youth and with colleagues), their perception of institutional climate, their relationship with themselves, and difficulties they might have felt during on using the strategies and contents learned on the MSC program. This data will be analysed through thematic, content, and discourse analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for caregivers:

Professionals working in YDC for at least 6 months Professionals that directly interacte with the delinquent youth on a regular basis (minimum of 30/hours per week).

* Inclusion criteria for youth:

Youth that entered the YDC at least 3 months before the study's onset (adjustment time); Aged between 14 and 18 YO; Know how to read/write and Portuguese language.

Exclusion Criteria:

- Exclusion criteria for youth: Cognitive impairment or diagnosis of a psychotic disorder; Remaining in YDC for less than 9 months.

-

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
The Self-Compassion Scale (SCS) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The SCS (original version (OV) Neff, 2003; Portuguese version (PV) Castilho & Pinto-Gouveia, 2012) consists of a 26-item scale that intends to assess levels of self-compassion. It is composed of six factors, threebeing positive (i.e., Self-kindness, Common humanity, and Mindfulness) and three being and focusing on a lack of self-compassion (i.e., Self-judgment, Isolation, and Over-identification). Items are rated on a 5-point Likert scale (1 - almost never to 5 - almost always). Previous research on SCS has shown good psychometric properties (Castilho & Pinto-Gouveia, 2012; Neff, 2003).
Compassion Scale (CS) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The CS (OV: Pommier, 2011; PV: Sousa et al., 2017) is a 24-item self-report questionnaire that measures compassion towards others and is composed of six subscales: Kindness; Common Humanity; Mindfulness; Indifference; Separation, and Disengagement. Items are rated using a five-point Likert scale (from 1 = almost never to 5 = almost always) according to how frequently participants feel and act towards others. Previous psychometric information showed good internal consistency values (Pommier, 2011; Sousa et al., 2017).
Fears of Compassion Scale (FCS) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The FCS (OV: Gilbert et al. 2011; PV: Simões, 2012) is a 38-item scale that comprises three subscales measuring: Fears of expressing compassion for others (composed of 10 items, 9 in the Portuguese version); Fears of receiving compassion from others; and Fears of expressing self-compassion (assessed for 15 items). The items are rated on a five-point Likert scale (0 = Do not agree at all to 4 = Completely agree). Previous psychometric studies reported very good internal consistency levels (Gilbert et al., 2011; Simões, 2012).
Cognitive and Affective Mindfulness Scale - Revised Form (CAMS-R) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The CAMS-R (OV: Feldman et al., 2007; PV: Teixeira & Pereira, 2015) consists of 12 itens intending to the degree to which individuals experience their thoughts and feelings and does not require meditation training. Items are answered on a 4-point Likert scale from 1 (not at all) to 4 (almost always). Previous research on CAMS-R reported acceptable to good internal consistency values (Feldman et al., 2007; Teixeira & Pereira, 2015).

SECONDARY OUTCOMES:
Professional Quality of Life Scale - version 5 (ProQOL-5) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The ProQOL-5 (OV: Stamm, 2009; PV: Carvalho, 2011) is a 30-item self-report measure composed of three subscales: Compassion Satisfaction, Burnout, and Secondary Traumatic Stress (STS). Items are rated on a 5-point Likert scale (from 1 = Never to 5 = Very Often), indicating how frequently each item was experienced by participants in the previous 30 days. Previous research on ProQOL-5 has shown good psychometric properties (Carvalho, 2011).
Depression, Anxiety, and Stress Scale - 21 (DASS-21) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The DASS-21 (OV: Lovibond & Lovibond, 1995; PV: Pais-Ribeiro et al., 2004) is a 21-item scale measuring Depression, Anxiety and Stress symptoms. Participants are asked to indicate the degree to which each statement applied to them in the last week, using a 4-point Likert scale (0 = Did not apply to me at all to 3 = Applied to me very much, or most of the time). Only the anxiety and depression subscales were used. Previous research on DASS-21 has shown good psychometric properties (Lovibond & Lovibond, 1995; PV: Pais-Ribeiro et al., 2004).
The Caring Shame and Guilt Scale (CSGS) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The CSGS (OV: Martin et al., 2006; PV: Salgueiro & Castilho, 2015) is a 12-item scale that assesses feelings of shame and guilt related to caring. Shame items focus on the key domains of shame relating to self-criticism, needing to live up to other people's expectations, and fear of criticism from others. Guilt items focus on fears of harming others, regret, and the sense of responsibility. Participants are instructed to respond to items on a 4-point Likert scale from 0 (not at all like me) to 4 (extremely like me). Previous research with university students reported very good results on internal consistency (Salgueiro & Castilho, 2015). This measure is currently being adapted and validated to two Portuguese samples of adult caregivers (i.e., caregivers of delinquent youth and parents of adolescents).
Social Connectedness Scale - Revised Form (SCS-R) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The SCS-R (OV: Lee et al., 2001; OV: Francisco, et al., 2011) measures the degree of interpersonal closeness that the individual experiences in their social world, including family, peers, friends, and society in general. This single-factor scale is composed of 20 items, 10 formulated in a positive form and 10 items in a negative way. Items are rated on a 6-point Likert scale (1 = strongly disagree; 6 = strongly agree). Previous research on SCS-R presented a very good internal consistency (Lee et al., 2001; Francisco, et al., 2011).
General Work-Related Stress Questionnaire (QSo-G) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The QSO-G (Gomes, 2010) assesses potential causes of work-related stress, and is divided into two parts: in the first part, participants are asked about the global level of stress that they feel related to their professional activity; the second part concerns potential sources of stress, divided into seven dimensions (i.e., relationship with the receptors of their services, with hierarchy superiors and with colleagues; overwork; career and payment; familiar issues and work material and human resources). All items are rated on a five-point Likert scale: 0=No stress; 2=Moderated Stress; 4=High Stress). Previous research reported acceptable internal consistency values (Gomes, 2010).
OSQ (Ocupational satisfaction questionnaire) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  The QSO (Freixo, 2010) is a 12-item self-report questionnaire aiming to assess specific criteria related to job satisfaction, based 3 factors: Perceived value given to ones' work; Safety and working conditions, and work-related interactions and work performance. Items are rated on a 6-point Likert scale about participants' satisfaction on those job issues (1= extremely unsatisfied to 6= extremely satisfied). QSO presented acceptable to good internal consistency values (Freixo, 2010).
World Health Organization Quality of Life-Brief (WHOQOL-BRIEF) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  WHOQOL-BREF (OV: WHOQOL Group, 1994 (World Health Organization Quality of Life Group; PV: Canavarro, et al., 2006) is a multidimensional and multicultural self-report measure that uses 26 itens to assess quality of life based on four dimensions: Physical; Psychological; Social Relationships, and Environment, rated on a 5-point Likert scale which varies according to the assessed dimension (1=Nothing/Very Bad/Very unsatisfied to 5=Completely/Very Good/Very satisfied). Previous research on WHOQOL-Brief has reported good to very good internal consistency indices (World Health Organization Quality of Life Group; Canavarro, et al., 2006).
Current Warmth and Safeness experiences (CEWSS-A) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will respond to the CEWSS-A (Santos, et al., 2020), which is a 12-item self-report measure designed to assess the frequency in which adolescents feel emotional experiences of warmth, care, and safety with others, in the period of the last two weeks. Items are answered using a Likert-scale response ranging from 0 (No, never) to 4 (Yes, most of the time). Previous research on CEWSS-A reported very good internal consistency indices (Santos et al., 2020).
Social Connectedness Scale - Revised Adolescents Form (SCS-RA) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will respond to the SCS-RA (OV: Lee et al., 2001; PV: Francisco, et al., 2011) that measures the degree of interpersonal closeness that the individual experiences in his or her social world, including family, peers, friends, and society in general. This single-factor scale is composed of 20 items, 10 formulated in a positive form and 10 items in a negative way. Items are rated on a 6-point Likert scale (1 = strongly disagree; 6 = strongly agree). Previous research on SCS-R presented a very good internal consistency (Lee et al., 2001; Francisco, et al., 2011). This measure was adapted and is currently being validated for two Portuguese samples of adolescents (i.e., a forensic and a community sample).
Other as Shamer - Brief Form for adolescents (OAS-BA) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will fulfil to the OAS-BA (Cunha et al., 2015), which is a short version of the Other as Shamer Scale (Goss et al., 1994). It inclused eight items to assesseexternal shame (i.e., the subject's perception of being negatively judged by others), rated on a 5-point scale, reporting how frequently one experiences the feelings described in each statement (0 = never to 4 = almost always). Previous research on OAS-BA showed good to very good internal consistency (Cunha et al., 2015; Sousa et al., 2022).
Self-Compassion Scale - Adolescent version (SCS-A) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will fulfil to the SCS-A (OV: Neff, 2003; PV for adolescents: Cunha et al., 2016) which is a 26-item scale assessing self-compassion and comprising six subscales:
  Self-kindness, Self-judgment, Common Humanity, Isolation, Mindfulness and Over-identification. Participants are asked to answer each item, related to the question "How I typically act towards myself in difficult times", using a 5-point scale (1 = Almost never; 5 = Almost Always). Previous research with adolescents presented a good to very internal consistency for the total score as well as for subscales (Cunha et al., 2016; Sousa et al., 2022).
KIDSSCREEN-27 | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will respond to the KIDSCREEN-27 (OV.:WHOQOL Group, 1994 (World Health Organization Quality of Life Group; pv: Gaspar & Gaspar de Matos, 2008) that is a reduced form of KIDESCREEN-52 which intends to understand and characterize the perception of youth about their quality of life, based on five dimensions: Physical Well-Being; Psychological Well-Being; Autonomy and Parent Relations; Peers and Social Support; School Environment, rated on a 5-point Likert scale (1= nothing to 5=totally). In this study, only Physical and Psychological Well-being and School Environment dimensions were used. Previous research on KIDESCREEN-27, has shown acceptable to good internal consistency indices (Gaspar & Gaspar de Matos, 2008).
Proposed Specifiers for Conduct Disorder (PSCD) | Baseline, Week 13, Follow-Up 3 Months and Follow-Up 6 Months
  Youth will respond to PSCD (Ribeiro da Silva et al., 2023) which is a 24-item psychopathic trait measure designed for administration in youths and addressing four subscales: grandiose-manipulative, callous-uncaring, daring-impulsive, and Conduct Disorder. Each factor is estimated by a set of six items, each rated on a 3-point Likert scale (0 = not true; 1 = somewhat true; 2 = true). Previous research on PSCD showed good internal consistency indicators for the total score and acceptable ones for the subscales (Ribeiro da Silva et al., 2023).

OTHER OUTCOMES:
Individual interviews for assessing qualitatively the perception of the impact of the MSC program | Follow-Up 3 Months and Follow-Up 6 Months
  In order to assess the participants' perception about their experience with the intervention, individual interviews (II) will be conducted 3 and 6 months after the final MSC session with the caregivers who attended the treatment group. The II will be composed of 4 to 8 open-ended questions, regarding the experiences and perception of impact/change on the caregivers' daily routine at the YDC, on the relationship with themselves and with others as also on difficulties related to the maintenance of the practices. The II will be audio-recorded and transcribed verbatim.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene M Paulo, Master, Principal Investigator — Faculty of Psychology and Educational Sciences - University of Coimbra.
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), Faculty of Psychology and Educational Sciences - University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baetz CL, Surko M, Moaveni M, McNair F, Bart A, Workman S, Tedeschi F, Havens J, Guo F, Quinlan C, Horwitz SM. Impact of a Trauma-Informed Intervention for Youth and Staff on Rates of Violence in Juvenile Detention Settings. J Interpers Violence. 2021 Sep;36(17-18):NP9463-NP9482. doi: 10.1177/0886260519857163. Epub 2019 Jun 28. PMID 31253054
- [Background] Cocker F, Joss N. Compassion Fatigue among Healthcare, Emergency and Community Service Workers: A Systematic Review. Int J Environ Res Public Health. 2016 Jun 22;13(6):618. doi: 10.3390/ijerph13060618. PMID 27338436
- [Background] Dev V, Fernando AT 3rd, Lim AG, Consedine NS. Does self-compassion mitigate the relationship between burnout and barriers to compassion? A cross-sectional quantitative study of 799 nurses. Int J Nurs Stud. 2018 May;81:81-88. doi: 10.1016/j.ijnurstu.2018.02.003. Epub 2018 Feb 21. PMID 29518624
- [Background] Dolitzsch C, Schmid M, Keller F, Besier T, Fegert JM, Schmeck K, Kolch M. Professional caregiver's knowledge of self-reported delinquency in an adolescent sample in Swiss youth welfare and juvenile justice institutions. Int J Law Psychiatry. 2016 Jul-Aug;47:10-7. doi: 10.1016/j.ijlp.2016.02.026. Epub 2016 Apr 3. PMID 27048623
- [Background] Duarte J, Pinto-Gouveia J. Effectiveness of a mindfulness-based intervention on oncology nurses' burnout and compassion fatigue symptoms: A non-randomized study. Int J Nurs Stud. 2016 Dec;64:98-107. doi: 10.1016/j.ijnurstu.2016.10.002. Epub 2016 Oct 8. PMID 27744228
- [Background] Faragher EB, Cass M, Cooper CL. The relationship between job satisfaction and health: a meta-analysis. Occup Environ Med. 2005 Feb;62(2):105-12. doi: 10.1136/oem.2002.006734. PMID 15657192
- [Background] Harder AT, Knorth EJ, Kalverboer ME. Risky or Needy? Dynamic Risk Factors and Delinquent Behavior of Adolescents in Secure Residential Youth Care. Int J Offender Ther Comp Criminol. 2015 Sep;59(10):1047-65. doi: 10.1177/0306624X14531036. Epub 2014 Apr 21. PMID 24752639
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Ribeiro da Silva D, Rijo D, Brazao N, Paulo M, Miguel R, Castilho P, Vagos P, Gilbert P, Salekin RT. The efficacy of the PSYCHOPATHY.COMP program in reducing psychopathic traits: A controlled trial with male detained youth. J Consult Clin Psychol. 2021 Jun;89(6):499-513. doi: 10.1037/ccp0000659. PMID 34264698
- [Background] Rijo D, Brazao N, Barroso R, da Silva DR, Vagos P, Vieira A, Lavado A, Macedo AM. Mental health problems in male young offenders in custodial versus community based-programs: implications for juvenile justice interventions. Child Adolesc Psychiatry Ment Health. 2016 Nov 1;10:40. doi: 10.1186/s13034-016-0131-6. eCollection 2016. PMID 27822300
- [Background] Rijo D, Miguel RR, Paulo M, Brazao N. The Effects of the Growing Pro-Social Program on Early Maladaptive Schemas and Schema-Related Emotions in Male Young Offenders: A Nonrandomized Trial. Int J Offender Ther Comp Criminol. 2020 Oct;64(13-14):1422-1442. doi: 10.1177/0306624X20912988. Epub 2020 Apr 10. PMID 32274945
- [Background] Sichel CE, Burson E, Javdani S, Godfrey EB. Theorizing Safety Informed Settings: Supporting Staff at Youth Residential Facilities. Am J Community Psychol. 2019 Jun;63(3-4):405-417. doi: 10.1002/ajcp.12307. Epub 2019 Feb 13. PMID 30758850
- [Background] Sinclair S, Kondejewski J, Raffin-Bouchal S, King-Shier KM, Singh P. Can Self-Compassion Promote Healthcare Provider Well-Being and Compassionate Care to Others? Results of a Systematic Review. Appl Psychol Health Well Being. 2017 Jul;9(2):168-206. doi: 10.1111/aphw.12086. Epub 2017 Apr 10. PMID 28393485
- [Background] Sinclair S, Raffin-Bouchal S, Venturato L, Mijovic-Kondejewski J, Smith-MacDonald L. Compassion fatigue: A meta-narrative review of the healthcare literature. Int J Nurs Stud. 2017 Apr;69:9-24. doi: 10.1016/j.ijnurstu.2017.01.003. Epub 2017 Jan 12. PMID 28119163
- [Background] Walden AL, Allen NE. Examining Correctional Staff Members' Engagement in Rehabilitation as Part of Their Everyday Practices in Short-term Juvenile Detention. Am J Community Psychol. 2019 Dec;64(3-4):310-320. doi: 10.1002/ajcp.12369. Epub 2019 Aug 2. PMID 31373031
- [Background] Bazzano, A., Wolfe, C., Zylowska, L., Wang, S., Shuster, E., Barret,C., & Lehrer, D. (2013). Mindfulness Based Stress Reduction (MBSR) for Parents and Caregivers of Individuals with Developmental Disabilities: A Community-Based Approach. Journal of Child and Family Studies, 24, 298-308. https://doi.org/10.1007/s10826-013-9836-9
- [Background] Barford, S.W. &Whelton, W. J. (2010). Understanding Burnout in Child and Youth Care Workers. Child Youth Care Forum, 39:271-287. https://doi.org/10.1007/s10566-010-
- [Background] Boellinghaus, I., Jones, F. W., & Hutton, J. (2012). The role of Mindfulness and Loving Kindness in Cultivating Self-Compassion and Other-Focused Concern in Health Care Professionals. Minfulness, 5, 129-138. https://doi.org/10.1007/s12671-012-0158-6
- [Background] Conboy, J. (2003). Algumas medidas típicas univariadas da magnitude do efeito. Análise Psicológica, 2(21), 145- 158. http://www.scielo.oces.ctes.pt/pdf/aps/v21n2/v21n2a02.pdf
- [Background] Cox, A. (2018). Juvenile Facility Staff Contestations of Change. Youth Justice, 18, 248-264. https://doi.org/10.1177/1473225418794104
- [Background] Harder, A. T., Knorth, E.J., & Kalverboer, M. E. (2013). A secure base? The adolescent-staff relationship in residential youth care. Child & Family Social Work, 18 (3), 305-317. https://doi.org/10.1111/j.1365-2206.2012.00846.x
- [Background] Jolivette, K., Swoszowski, N. C., Kumm, S., Sanders, S., & Ansley, B. M. (2019). Embedding Staff Self-Care into the MTSS Framework for Those Working in Juvenile Correctional Facilities. Journal of Correctional Education, 70(1), 2-19. https://doi.org/10.1177/0741932519880336
- [Background] Kabat-Zinn, J. (1990). Full Catastrophe Living: Using the Wisdom of Your Body and Mind to Face Stress, Pain and Illness. Dell.
- [Background] Lary, D. (2007).The effect of educational Program for Direct care workers on attitude of stigma toward mentally ill youth in a Juvenile Justice System. Dissertation presented to the Graduate Faculty in Partial Fulfillment of the Requirements for the Degree of Doctor of Nursing Science. New Orleans, Louisiana State University Health Sciences Center School of Nursing.
- [Background] Mathys, C. (2017). Effective components of interventions in juvenile justice facilities: How to take care of delinquent youths? Children and Youth Services, 73, 319-327. https://doi.org/10.1016/j.childyouth.2017.01.007
- [Background] Newsome, S., Waldo, M., & Gruska, C. (2012). Mindfulness Group Work: Preventing Stress and Increasing Self-Compassion Among Helping Professionals in Training. The Journal for Specialists in Group Work, 37(4), 297-311. https://doi.org/10.1080/01933922.2012.690832
- [Background] Wilson, A. C., Mackintosh, K., Power, K., & Chan, S. W. Y. (2018). Effectiveness of Self-Compassion Related Therapies: A Systematic Review and Meta-analysis. Mindfulness, 1-17. https://doi.org/10.1007/s12671-018-1037-6
- [Background] Canavarro, M. C., Simões, M. R., Vaz Serra, A., Pereira, M., Rijo, D., Quartilho, M. J., ... Carona, C. (2007). Instrumento de avaliação da qualidade de vida da Organização Mundial de Saúde: WHOQOL-Bref. In M. Simões, C. Machado, M. Gonçalves, & L. Almeida (Eds.), Avaliação psicológica: Instrumentos validados para a população portuguesa (Vol. III, pp. 77-100). Quarteto Editora.
- [Background] Carvalho, P. (2011). Estudo da fadiga por compaixão nos cuidados paliativos em Portugal: Tradução e adaptação cultural da escala "Professional Quality of Life 5. Unpublished Master Thesis. Universidade Católica Portuguesa, Porto.
- [Background] Castilho, P., & Pinto-Gouveia, J. (2011). Autocompaixão: Estudo da validação da versão portuguesa da Escala da Autocompaixão e da sua relação com as experiências adversas na infância, a comparação social e a psicopatologia [self-compassion: Validation study of the Portuguese version of Self-compassion and their relation with adverse experiences in Childhood, social comparison, and psychopathology]. Psychologica, 54, 203-231.
- [Background] Cunha, M., Xavier, A., & Castilho, P. (2016). Understanding self-compassion in adolescents: Validation study of the Self-Compassion Scale. Personality and Individual Differences, 93, 56-62. https://doi.org/10.1016/j.paid.2015.09.023
- [Background] Cunha, M., Xavier, A., Cherpe, S., & Pinto-Gouveia, J. (2015). Avaliação da Vergonha em Adolescentes: "The Other as Shamer Scale". Psicologia: Teoria e Pesquisa (Brasília), 33, 1-19. https://doi.org/10.1590/0102.3772e3336
- [Background] Feldman, G. C., Hayes, A. M., Kumar, S. M., Greeson, J. M., & Laurenceau, J. P. (2007). Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness Scale---Revised (CAMS-R). Journal of Psychopathology and Behavioral Assessment, 29, 177---190. http://dx.doi.org/10.1007/s10862-006-9035-8
- [Background] Francisco, R., Crespo, C., Dias, E., Malaquias, A. S. & Rocha, I. (2011). Versão portuguesa da SCS-R (versão para investigação). Universidade de Lisboa, Lisboa.
- [Background] Freixo, L. (2010). Das fontes de satisfação no trabalho organizacional: Estudo em duas empresas do setor metalúrgico do Norte do País. Tese de Metrado apresentada à Faculdade de Ciências Humanas e Sociais da Universidade Fernando Pessoa no Porto.
- [Background] Gilbert P, McEwan K, Matos M, Rivis A. Fears of compassion: development of three self-report measures. Psychol Psychother. 2011 Sep;84(3):239-55. doi: 10.1348/147608310X526511. Epub 2011 Apr 13. PMID 22903867
- [Background] Gomes, A.R. (2010). Questionário de Stresse Ocupacional - Versão Geral (QSO-VG). Relatório técnico não publicado. Braga: Universidade do Minho.
- [Background] Lee, R. M., Draper, M., & Lee, S. (2001). Social connectedness, dysfunctional interpersonal behaviors, and psychological distress: Testing a mediator model. Journal of Counseling Psychology, 48(3), 310-318. https://doi.org/10.1037/0022-0167.48.3.310
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Martin Y, Gilbert P, McEwan K, Irons C. The relation of entrapment, shame and guilt to depression, in carers of people with dementia. Aging Ment Health. 2006 Mar;10(2):101-6. doi: 10.1080/13607860500311953. PMID 16517484
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2(3), 223-250. https://doi.org/10.1080/15298860309027
- [Background] Pais-Ribeiro, J. L., Honrado, A., & Leal, I. (2004). Contribuição para o estudo da adaptação portuguesa das escalas de ansiedade, depressão e stress (EADS) de 21 itens de Lovibond e Lovibond. Psicologia, Saúde e Doenças, 5(1), 229-239.
- [Background] Pommier, E. A. (2010). The compassion scale [Doctoral dissertation, The University of Texas at Austin]. https://repositories.lib.utexas.edu/handle/2152/ETD-UT-2010-12-2213
- [Background] Ribeiro da Silva D, Sousa R, Rijo D, Mendez B, Tsang S, Salekin RT. Proposed Specifiers for Conduct Disorder (PSCD): Factor Structure and Validation of the Self-Report Version in Community and Forensic Samples of Portuguese Youth. Assessment. 2023 Jan;30(1):124-143. doi: 10.1177/10731911211044534. Epub 2021 Sep 15. PMID 34523369
- [Background] Salgueiro, A., & Castilho, P. (2015). As emoções autoconscientes e o papel do cuidador: análise fatorial confirmatória e propriedades psicométricas da versão portuguesa da Escala de Vergonha e Culpa no Cuidar (EVCC) [Tese de Mestrado]. Universidade de Coimbra.
- [Background] Santos L, Sousa R, Pinheiro MDR, Rijo D. Development and Validation of the Current Experiences of Warmth and Safeness Scale in Community and Residential Care Adolescents. Child Psychiatry Hum Dev. 2021 Dec;52(6):1118-1130. doi: 10.1007/s10578-020-01090-6. Epub 2020 Nov 1. PMID 33130924
- [Background] Simões, D. (2012). Medo da Compaixão: estudo das propriedades psicométricas da Fears of Compassion Scales (FCS) e estudo da sua relação com medidas de Vergonha, Compaixão e Psicopatologia. Dissertação de Mestrado apresentada à Faculdade de Psicologia e Ciências da Educação da Universidade de Coimbra. http://hdl.handle.net/10316/23280
- [Background] Sousa, R., Castilho, P., Vieira, C., Vagos, P., & Rijo, D. (2017). Dimensionality and gender-based measurement invariance of the Compassion Scale in a community sample. Personality and Individual Differences, 117, 182-187. https://doi.org/10.1016/j.paid.2017.06.003
- [Background] Sousa R, Paulo M, Brazao N, Castilho P, Rijo D. Measuring compassion toward others: Dimensionality of the compassion scale in community adolescents and in adolescents with behavioral disorders. Psychol Assess. 2022 Jul;34(7):631-642. doi: 10.1037/pas0001133. Epub 2022 Mar 31. PMID 35357875
- [Background] Stamm, B. H. (2009). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL). Retrived from www.proqol.org Stamm, B. H. (2009). Professional Quality of Life: Compassion Satisfaction and Fatigue Version 5 (ProQOL).
- [Background] Teixeira, R., Ferreira, G., & Pereira, M. G. (2017) Portuguese validation of the Cognitive and Affective Mindfulness Scale-Revised and the Philadelphia Mindfulness Scale. Mindfulness & Compassion, 2, 3-8. http://dx.doi.org/10.1016/j.mincom.2017.03.001
- [Background] The WHOQOL Group. (1994). Development of the WHOQOL: Rationale and current status. International Journal of Mental Health, 23(3), 24-56.